CLINICAL TRIAL: NCT03384628
Title: An Evaluation Of The Fitting Success Rate Of Senofilcon A Soft Contact Lenses In Three Designs.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Graeme Young (Other)
Collaborators: Visioncare Research Ltd. (Other)
Responsible Party: Sponsor-Investigator, Graeme Young, Graeme Young PhD MPhil FCOptom DCLP, Visioncare Research Ltd.
Organization: Visioncare Research Ltd. (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TRTN-501
Record Dates: First submitted 2017-12-08; First posted 2017-12-27 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-04

CONDITIONS: Myopia
Keywords: Contact lens; The Young Theory
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Each subject will wear the three contact lens types bilaterally in random succession
Who Masked: Participant
Masking Description: Subjects will be masked to lens type and lens codes. A sealed decoding envelope will be provided to the investigator. In the event of an emergency the investigator will break the masking and the medical monitor will be notified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- First Pair Senofilcon A contact lens (Active Comparator): The first pair of Senofilcon A contact lenses is applied (according to the fitting schedule), allowed to settle before assessment of the first pair Senofilcon A contact lens and subsequent removal.
  Interventions: Device: First pair Senofilcon A contact lens
- Second pair Senofilcon A contact lens (Active Comparator): The second pair of contact lenses is applied (according to the fitting schedule), allowed to settle before assessment of the second pair Senofilcon A contact lens and subsequent removal.
  Interventions: Device: Second pair Senofilcon A contact lens
- Third pair Senofilcon A contact lens (Active Comparator): The third pair of Senofilcon A contact lens is applied (according to the fitting schedule), allowed to settle before assessment of the third pair Senofilcon A contact lens and subsequent removal.
  Interventions: Device: Third pair Senofilcon A contact lens

INTERVENTIONS:
Device: First pair Senofilcon A contact lens — Fit assessment of the first pair contact lenses.
  Arms: First Pair Senofilcon A contact lens
Device: Second pair Senofilcon A contact lens — Fit assessment of the second pair of contact lenses.
  Arms: Second pair Senofilcon A contact lens
Device: Third pair Senofilcon A contact lens — Fit assessment of the third pair of contact lenses.
  Arms: Third pair Senofilcon A contact lens

SUMMARY:
This study will compare the on-eye fitting characteristics of three types of contact lenses. Each lens pair will be worn for 30 to 45 minutes before assessment and the results will be compared to mathematically calculated fitting characteristics.

DETAILED DESCRIPTION:
This will be an approx. 40-60 subject, one-day, double-masked, randomised, repeated measures study. Each subject will wear the three lens types bilaterally in random succession, a total of six lenses will therefore be worn by each subject (3 per eye).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years.
* Able to read, comprehend and sign an informed consent.
* Willing to comply with the wear and study assessment schedule.
* Spherical distance prescription between -0.50 and -6.00 (inc.).
* Astigmatism, if present,≤1.50DC in both eyes.
* Have normal eyes with no evidence of any ocular abnormality or disease. For the purposes of this study a normal eye is defined as one having:

A clear central cornea. No anterior segment disorders. No clinically significant slit lamp findings (i.e. corneal oedema, significant staining, central scarring, infiltrates, active neovascularisation). No other active ocular disease (including pterygia).

Exclusion Criteria:

* Previous anterior ocular surgery
* Any active corneal infection, injury or inflammation

  . •Large pinguecula likely to affect soft lens fit
* Systemic or ocular disease or medication which might interfere with CL wear
* Pregnancy or breastfeeding
* Participation in any concurrent trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Lens fit (position on the eye) in mm | 25 minutes
  Horizontal Lens Centration (mm), Vertical Lens Centration (mm), Post-blink movement in primary gaze (mm), Version lag (mm), Horizontal corneal overlap (mm), Diameter acceptance (mm),
Lens edge tightness fit grade 0-4 | 5 minutes
  Edge tightness (grade 0-4)
Lens tightness fit graded as % | 5 minutes
  Tightness (push-up %),
Lens overall fit grade 0-5 | 5 minutes
  Overall fit acceptability (Grade 0-5),

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Young, PhD MPhil, Study Director — Managing director
Locations (2):
- United Kingdom (2):
  - Visioncare research, Farnham, Surrey
  - Aston University Optometry Clinic, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT03384628/Prot_000.pdf
  • Informed Consent Form (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT03384628/ICF_001.pdf
  • Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT03384628/SAP_002.pdf